CLINICAL TRIAL: NCT00823875
Title: A Randomized, Control, Open Label, Multicentre Clinical Study to Evaluate the Efficacy and Safety of Cilostazol and Probucol Alone and in Combination on Atherosclerosis Related Biomarker---atherosclerosis Cerebral Infarction Patient as Study Subject
Brief Title: Study of Cilostazol and Probucol Alone and in Combination on Atherosclerosis Related Biomarker---atherosclerosis Cerebral Infarction Patient as Study Subject
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Quanjie Wei, Otsuka Beijing Research Institue
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 260-08-803-01
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-01

CONDITIONS: Atherosclerosis Cerebral Infarction
MeSH Terms: interventions — Cilostazol; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Cilostazol group
- 2 (Experimental)
  Interventions: Drug: Probucol group
- 3 (Experimental)
  Interventions: Drug: Cilostazol + Probucol group
- 4 (Other): Control Group
  Interventions: Drug: control group

INTERVENTIONS:
Drug: Cilostazol group — Cilostazol: At first, 50 mg (1 tablets) Bid, PO after breakfast and dinner. After administration of study drug for 1 week, and if patient has no significant discomfort, the drug dosage will increase to 100mg（2 tablets）Bid.
  Other Names: Pletaal
  Arms: 1
Drug: Probucol group — Probucol: 250 mg (1 tablet) Bid, PO after breakfast and dinner
  Other Names: Changtai
  Arms: 2
Drug: Cilostazol + Probucol group — Cilostazol: At first, 50 mg (1 tablets) Bid, PO after breakfast and dinner. After administration of study drug for 1 week, and if patient has no significant discomfort, the drug dosage will increase to 100mg（2 tablets）Bid.
  Probucol: 250 mg (1 tablet) Bid, PO after breakfast and dinner
  Other Names: Pletaal and Changtai
  Arms: 3
Drug: control group — routine treatment
  Other Names: Routine Treatment
  Arms: 4

SUMMARY:
Randomized, control, open label, multicentre clinical study. The patient who are in accordance with subject inclusion and exclusion criteria will be randomized to A group: Routine treatment B group: Routine treatment+ Cilostazol; C group : Routine treatment + Probucol; D group: Routine treatment+ Cilostazol+ Probucol .

DETAILED DESCRIPTION:
Efficacy index:

After 12 weeks of treatment, the change difference of arteriosclerosis related biomarker between 4 modality groups.

Pharmacokinetics:

After 12 weeks of treatment, the study medication plasma concentration including of Probucol ,Cilostazol , Cilostazol metabolism OPC-13015 and OPC-13213 will be measured.

Safety evaluation:

Analysis the abnormality of Adverse Event, Vital Sign, Physical Examination, 12-lead ECG, and Laboratory Tests (including blood routine examination, routine urine analysis, blood biochemistry examination, glycosylated hemoglobin) in 4 modality groups.

ELIGIBILITY:
Inclusion Criteria:

1. 40～80-year-old male or female
2. By brain CT or MRI result, cerebral infarction is clarified diagnosis within 1 year
3. With atherosclerosis, atherosclerosis should meet at least one of the conditions as below:

   * Clarified diagnosis of type 2 diabetes before
   * Clarified diagnosis of primary hypertension before
   * Clarified diagnosis of Atherosclerotic stenosis in any 2 or more than 2 regions as cerebral artery, carotid, extremity artery and coronary by conformation of ultrasonic or angiography result
4. Has Aspirin regularly for more than 1 month before registration
5. Informed Consent Form signature

Exclusion criteria：

1. Has an allergic history to study drugs( including of Probucol and Cilostazol) and Aspirin
2. Had lipid-lowing agents within the last 3 months ( except Statins)
3. Had antiplatelet or anticoagulation agents within the last 3 months (except Aspirin)
4. Had acute cerebral infarction within the last 1 month
5. Has cardiogenic cerebral embolism
6. At the registration ,Modified Rankin Scale ≥ 4
7. Hemorrhagic tendency or hemorrhagic disease (such as cerebral hemorrhage, gastrointestinal tract hemorrhage, etc.)
8. Had a myocardial infarction, angina pectoris within the last 3 months
9. Congestive heart failure
10. Is pregnant, is potentially pregnant, or is breastfeeding
11. Severe hepatic inadequacy or severe renal inadequacy (AST or ALT is 2.5 times higher than the upper limit of the normal value range, or serum creatinine is 1.2 times higher than the upper limit of the normal value range)
12. Persistent or hardly controlled hypertension (such as malignant hypertension, BP> 160/100 mmHg)
13. Severe ventricular arrhythmia (such as multiple and multifocal premature ventricular contractions)
14. Has a medical history that includes a cardiac syncope or a primary syncope
15. Has a condition that may prolong QT interval (such as congenital long QT syndrome, taking drugs which prolong QT interval, hypokalemia or hypomagnesemia, etc.)
16. Has severe diseases (such as, malignant tumor, severe anaemia, severe hematologic diabetes mellitus ketoacidosis, nonketotic hyperosmolar diabetic coma, etc.)
17. Registered other clinical trails within the last 3 months
18. Has vasculitis, moyamoya disease and other non-atherosclerosis vascular diseases
19. Other conditions that could exclude the subject from this study by doctor's judgment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
After 12 weeks of treatment, the change difference of arteriosclerosis related biomarker between 4 modality groups. | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Yining Huang, M.D., Principal Investigator — Peking University First Hospital
Locations (1):
- First Affliate Hospital of Beijing University, Beijing, China